CLINICAL TRIAL: NCT06073821
Title: A Phase 3, Open-Label, Randomized Study of Sonrotoclax (BGB-11417) Plus Zanubrutinib (BGB-3111) Compared With Venetoclax Plus Obinutuzumab in Patients With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Study of Sonrotoclax (BGB-11417) Plus Zanubrutinib (BGB-3111) Compared With Venetoclax Plus Obinutuzumab in Participants With Chronic Lymphocytic Leukemia (CLL)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-301; CTR20241195 (Other: ChinaDrugTrials)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-06

CONDITIONS: CLL
Keywords: CLL; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sonrotoclax Plus Zanubrutinib (Experimental): Participants will receive from start of Cycle 1 a standard dose of zanubrutinib once or twice daily orally and in combination with sonrotoclax starting from Cycle 4 onwards at increasing doses until target dose is reached and continuing until end of Cycle 15 (each cycle is 28 days)
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib
- Venetoclax Plus Obinutuzumab (Active Comparator): Participants will receive obinutuzumab 100mg intravenously on Day 1 Cycle 1, followed by 900 mg on Day 2 Cycle 1 (or alternatively receive 1000 mg intravenously on Day 1), followed by 1000 mg on Days 8 and 15 of Cycle 1 and thereafter on Day 1 of Cycles 2 through 6 (each cycle is 28 days) in combination with venetoclax at increasing doses until target dose is reached from Day 22 Cycle 1 until end of Cycle 12 (each cycles is 28 days)
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Sonrotoclax — Administered orally
  Other Names: BGB-11417
  Arms: Sonrotoclax Plus Zanubrutinib
Drug: Zanubrutinib — Administered orally
  Other Names: BGB-3111
  Arms: Sonrotoclax Plus Zanubrutinib
Drug: Venetoclax — Administered orally
  Arms: Venetoclax Plus Obinutuzumab
Drug: Obinutuzumab — Administered intravenously
  Arms: Venetoclax Plus Obinutuzumab

SUMMARY:
The main objective of this study is to compare the efficacy of sonrotoclax plus zanubrutinib versus venetoclax plus obinutuzumab in participants with chronic lymphocytic leukemia (CLL)

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia is a type of blood cancer that affects people around the world. People with CLL suffer from enlarged lymph nodes, spleen, or liver, or have symptoms like night sweats, weight loss and fever. They have shorter life expectancy compared to healthy people. There is an urgent need for new treatment to prolong life and control disease-related symptoms.

In this study, participants with CLL without prior treatment will receive either venetoclax plus obinutuzumab combination treatment that is considered a standard first line treatment or receive sonrotoclax plus zanubrutinib. It is hypothesized that sonrotoclax plus zanubrutinib may be better than venetoclax plus obinutuzumab in treating CLL.

The main purpose of this study is to compare the duration the participants live without the CLL getting worse between participants who received sonrotoclax plus zanubrutinib versus venetoclax plus obinutuzumab. Approximately 652 participants will be included in this study around the world. Participants will have equal chance to be allocated to receive either of the treatment combinations.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve (TN) adults with confirmed diagnosis of CLL which requires treatment
* Eastern Cooperative Oncology Group (ECOG) score 0, 1, or 2
* Measurable disease by Computer Tomography/Magnetic Resonance Imaging
* Adequate liver function as indicated by aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x the institutional upper limits of normal (ULNs) value; serum total bilirubin < 3.0 x ULN
* Adequate renal function as defined as creatinine clearance ≥ 50 milliliters per minute

Exclusion Criteria:

* Previous systemic treatment for CLL
* Known prolymphocytic leukemia or history of, or currently suspected, Richter's transformation
* Known central nervous system involvement
* History of confirmed progressive multifocal leukoencephalopathy (PML)
* Uncontrolled hypertension

Note: Other protocol defined criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2032-02 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Progression Free Survival (PFS） | Up to approximately 9 years
  PFS is defined as the time from the date of enrollment to the date of first confirmed disease progression or death due to any cause, whichever occurs first, as determined by independent review committee (IRC)
Cohort 1: Rate of Undetectable Measurable Residual Disease | Up to one and a half years
  Undetectable measurable residual disease uMRD4 rate at the first Post- Treatment Follow-up (PTFU 1) Visit will be based on next-generation sequencing.

SECONDARY OUTCOMES:
Cohort 1: Complete Response Rate (CRR ) by IRC | Up to approximately 9 years
  CRR is defined as the percentage of participants that achieved best response of complete response (CR)/ complete response with incomplete hematopoietic recovery (CRi), determined by IRC.
Cohort 1: Overall Survival (OS) | Up to approximately 9 years
  OS is defined as time from the date of enrollment to the date of death because of any cause
Cohort 1: PFS by Investigator Assessment | Up to approximately 9 years
  PFS is defined as the time from the date of enrollment to the date of first confirmed disease progression or death due to any cause, whichever occurs first, as determined by investigator assessment
Cohort 1: CRR by Investigator Assessment | Up to approximately 9 years
  CRR is defined as the percentage of participants that achieved best response of complete response (CR)/ complete response with incomplete hematopoietic recovery (CRi), determined by Investigator Assessment
Cohort 1: Rate of Undetectable Measurable Residual Disease | Up to approximately 9 years
  The overall uMRD4 rate is defined as the percentage of participants who achieve uMRD status in peripheral blood before disease progression or start of new anti-CLL treatment (whichever is earlier), based on flow cytometry.
Cohort 1: Overall Response Rate (ORR) by IRC and Investigator Assessment | Up to approximately 9 years
  ORR is defined as the percentage of participants who achieve a response (CR, CRi, nodular partial remission (nPR), partial response (PR), and partial response with lymphocytosis [PR-L]), before disease progression or start of new anti-CLL treatment (whichever is earlier).
Cohort 1: Duration of Response (DOR) by IRC and Investigator Assessment | Up to approximately 9 years
  DOR is defined as the time from first qualifying response PR, PR-L, CR, or CRi) until CLL progression or death.
Pooled Cohorts: PFS by IRC and Investigator Assessment | Up to approximately 9 years
  PFS is defined as the time from the date of enrollment to the date of first confirmed disease progression or death due to any cause, whichever occurs first, as determined by IRC
Pooled Cohorts: ORR by IRC and Investigator Assessment | Up to approximately 9 years
  ORR is defined as the percentage of participants who achieve a response (CR, CRi, nodular partial remission (nPR), partial response (PR), and partial response with lymphocytosis [PR-L]), before disease progression or start of new anti-CLL treatment （whichever is earlier）.
Pooled Cohorts: DOR by IRC and Investigator Assessment | Up to approximately 9 years
  DOR is defined as the time from first qualifying response PR, PR-L, CR, or CRi) until CLL progression or death.
Pooled Cohorts: Rate of Undetectable Measurable Residual Disease | Up to approximately 9 years
  The overall uMRD4 rate is defined as the percentage of participants who achieve uMRD status in peripheral blood before disease progression or start of new anti-CLL treatment (whichever is earlier),based on next-generation sequencing.
Pooled Cohorts: CRR by IRC and Investigator Assessment | Up to approximately 9 years
  CRR is defined as the percentage of participants that achieved best response of complete response (CR)/ complete response with incomplete hematopoietic recovery (CRi), determined by Investigator Assessment
Cohort 1 and Pooled Cohorts: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to one and a half years for Sonrotoclax Plus Zanubrutinib group and 13 months for Venetoclax Plus Obinutuzumab group]
  Safety will be assessed by monitoring and recording of all treatment emergent adverse events (AEs) graded by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Cohort 1 and Pooled Cohorts: Change from baseline in European Organization for Research and Treatment of Cancer Quality of Life Cancer Questionnaire -Core 30 (EORTC QLQ-C30) Global Health Status/QoL (GHS) and Physical Functioning Scales | Every three cycles during the treatment period
  The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 =Not at all (best) to 4 =Very Much (worst) and 2 questions answered on a 7-point scale where 1 =Very poor (worst) to 7 =Excellent (best). Higher scores in GHS and functional scales indicate better quality of life.
Cohort 1 and Pooled Cohorts: Change from baseline in EORTC Quality of Life Questionnaire - Chronic Lymphocytic Leukemia Module 17 Items (QLQ-CLL17) Symptom Burden and Physical Condition Scales | Every three cycles during the treatment period
  The symptom burden and physical condition/fatigue will be measured by EQ-5D-5L. EQ-5D-5L is a standardized instrument that measures health-related quality of life for men with prostate cancer. EQ-5D consists of EQ-5D descriptive system and EQ visual analogue scale (VAS). EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Number of participants with various responses to the mobility questionnaire are reported.
Cohort 1 and Pooled Cohorts: Change from baseline in European Quality of Life 5-Dimensions 5-Levels Health Questionnaire （EQ-5D-5L) Visual Analogue Scale (VAS). | Every three cycles during the treatment period
  Mean change from baseline in EQ-5D-5L VAS. The EQ-5D-5L measures health outcomes using a VAS to record a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine. A higher score indicates better health outcomes.

CONTACTS AND LOCATIONS:
Locations (202):
- United States (40):
  - Alaska Oncology and Hematology, Llc, Anchorage, Alaska
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego (Ucsd) Moores Cancer Center, La Jolla, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - UCLA Department of Medicine Hematologyoncology, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Medicine, Palo Alto, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Northwestern University, Chicago, Illinois
  - Illinois Cancercare, Pc, Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mission Cancer and Blood, Waukee, Iowa
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute Pavilion, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - Clinical Research Alliance, Inc, Westbury, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Levine Cancer Institute (Lci), Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute At Ohio State University, Columbus, Ohio
  - Oncology Associates of Oregon Willamette Valley Cancer Center, Eugene, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Scri Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Institute, Richmond, Virginia
  - Vcu Health Systemmassey Comprehensive Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Gunderson Health System, La Crosse, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (12):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Genesiscare North Shore, St Leonards, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford PK, South Australia
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern East, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
- Austria (3):
  - Medizinische Universitatsklinik Innsbruck, Innsbruck
  - Universitatsklinik Fur Innere Medizin Iii Universitatsklinikum Der Pmu Landeskrankenhaus Salzburg, Salzburg
  - Hanusch Krankenhaus, Vienna
- Brazil (6):
  - Unesp Faculdade de Medicina Da Universidade Estadual Paulista Campus Botucatu, Botucatu
  - Hospital Erasto Gaertner, Curitiba
  - Centro Gaucho Integrado de Oncologia Hospital Mae de Deus, Porto Alegre
  - Hospital Das Clinicas Da Faculdade de Medicina de Ribeirao Preto Usp, Ribeirão Preto
  - Hcfmusp Servico de Hematologia, Hemoterapia E Terapia Celular, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Canada (11):
  - Arthur Je Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency the Vancouver Centre, Vancouver, British Columbia
  - Cancercare Manitoba, Winnipeg, Manitoba
  - Lakeridge Health, Oshawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Integre de Sante Et de Services Sociaux de La Monteregie Centre, Greenfield Park, Quebec
  - Centre Hospitalier de Luniversite de Montreal (Chum), Montreal, Quebec
  - Unite de Recherche Clinique Du Cisss Des Laurentides, SaintJerome, Quebec
  - Ciusss de Lestrie Chus, Sherbrooke, Quebec
  - Chu de Quebec Universite Laval, Hopital de Lenfant Jesus, Centre Integre de Cancerologie (Cic), Québec
- China (26):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Jieyang Peoples Hospital (Jieyang Affiliated Hospital, Sun Yat Sen University ), Jieyang, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Nanyang Central Hospital, Nanyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central Peoples Hospitaljiangnan Branch, Yichang, Hubei
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Jining No Peoples Hospital West Branch, Jining, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Czechia (6):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni Nemocnice Plzen, PLZE
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- France (13):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Chu Clermont Ferrand Therapie Cellulaire and Hematolo, Clermontferrand
  - Clinique Louis Pasteur, Esseylesnancy
  - Centre Hospitalier Le Mans, Le Mans
  - Chu Lille, Lille
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Hopital Prive Du Confluent, Nantes
  - Hopital de La Pitie Salpetriere, Paris
  - Chu Rennes, Rennes Cedes
  - Centre Henri Becquerel, Rouen
  - Chu Tours Hopital Bretonneau, Tours
  - Chu Nancy Hopital Brabois, VandoeuvrelesNancy
- Germany (3):
  - Praxis Am Volkspark, Berlin
  - Centrum Fur Haematologie Und Onkologie Bethanien, Frankfurt am Main
  - Universitaetsklinikum Schleswig Holstein Campus Luebeck, Lübeck
- Israel (5):
  - Assuta Ashdod Medical Center, Ashdod
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Assuta Medical Center, Tel Aviv
- Italy (7):
  - Azienda Ospedaliera Universitaria Policlinico Santorsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Di Ferrara, Ferrara
  - Istituto Europeo Di Oncologia, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Aou Maggiore Della Carita, Novara
  - Azienda Ospedaliera Di Padova, Padua
  - Ospedale Santa Maria Della Misericordia, Perugia
- Japan (19):
  - Aichi Cancer Center Hospital Clinical Oncology, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - Nho Shikoku Cancer Center, Matsuyama, Ehime
  - Aiiku Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center, AmagasakiCity, Hyōgo
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Tokai University Hospital, Iseharashi, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Kurashiki Central Hospital, Kurashikishi, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Sakai, Osaka
  - National Cancer Center Hospital, ChuoKu, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - Aomori Prefectural Central Hospital, Aomori
  - Kumamoto University Hospital, Kumamoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Yokohama Municipal Citizens Hospital, Yokohama
- Netherlands (9):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Amsterdam Umc Vu Mc, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Martini Ziekenhuis, Groningen
  - Ikazia Ziekenhuis, Rotterdam
  - Franciscus Gasthuis and Vlietland, Schiedam
  - Hagaziekenhuis, Sgravenhage
- New Zealand (6):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Tauranga Hospital, Tauranga
  - Wellington Regional Hospital (Ccdhb), Wellington
- Poland (6):
  - Wielospecjalistyczne Centrum Onkologii I Traumatologii Im M Kopernika W Lodzi, Lodz
  - Uniwersytecki Szpital Kliniczny Nr W Lublinie, Lublin
  - Uniwersytecki Szpital Kliniczny W Poznaniu, Poznan
  - Centralny Szpital Kliniczny Uck Wum, Warsaw
  - Instytut Hematologii I Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny Im Jana Mikulicza Radeckiego We Wroclawiu, Wroclaw
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- South Korea (6):
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - National Cancer Center (Korea), IlsandongGu GoyangSi, Gyeonggi-do
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
- Spain (8):
  - Hospital Universitario de Burgos, Burgos
  - Institut Catala Doncologia Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario de Gran Canaria Dr Negrin, Las Palmas de Gran Canaria
  - Md Anderson Cancer Center Madrid Spain, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital La Candelaria, Santa Cruz de Tenerife
- Karolinska Universitetssjukhuset Solna, Stockholm, Sweden
- Turkey (Türkiye) (4):
  - Ankara University Medical Faculty, Ankara
  - Gazi University, Ankara
  - Erciyes University School of Medicine, Kayseri
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
- United Kingdom (10):
  - University Hospitals Dorset Royal Bournemouth Hospital, Bournemouth
  - Kent and Canterbury Hospital, Canterbury
  - Churchill Hospital Oxford University Hospital Nhs Trust, Headington
  - St Jamess University Hospital, Leeds
  - The Clatterbridge Cancer Centre Liverpool, Liverpool
  - University College Hospital, London
  - Kings College, London
  - Norfolk and Norwich University Hospitals Nhs Foundation Trust, Norwich
  - Southampton General Hospital, Southampton
  - Royal Marsden Nhs Foundation Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/